CLINICAL TRIAL: NCT00410254
Title: An Open Label, Single-Dose Midazolam, Multiple-Dose HCV-796, Sequential 3-Period Study to Determine the Pharmacokinetics of the Potential Drug Interaction Between HCV-796 and Midazolam
Brief Title: HCV-796 and Midazolam Drug Interaction Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3173A1-109
Record Dates: First submitted 2006-12-08; First posted 2006-12-12 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Healthy
MeSH Terms: interventions — HCV 796; Midazolam

INTERVENTIONS:
Drug: HCV-796
Drug: midazolam

SUMMARY:
To evaluate the potential PK interaction of multiple oral doses of HCV-796 and a single oral dose of midazolam when coadministered to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and 12-lead ECG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2007-06; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Safety PK

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- United States (2):
  - Gainesville, Florida
  - Philadelphia, Pennsylvania